CLINICAL TRIAL: NCT00125437
Title: Safety and Efficacy of Larger Dose of Spironolactone for the Treatment of Patients With Nonischemic Cardiomyopathy
Brief Title: Larger Dose of Spironolactone for the Treatment of Patients With Nonischemic Cardiomyopathy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Poor compliance with the therapy and lot of patients were lost to follow up.
Sponsor: Hebei Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 05276101D-84
Record Dates: First submitted 2005-07-29; First posted 2005-08-01 (Estimated); Last update posted 2009-07-15 (Estimated); Status verified 2008-12

CONDITIONS: Heart Failure, Congestive
Keywords: aldosterone antagonists; spironolactone; left ventricular remodeling
MeSH Terms: conditions — Heart Failure; Ventricular Remodeling | interventions — Spironolactone

INTERVENTIONS:
Drug: spironolactone

SUMMARY:
The purpose of this study is to determine whether a larger dose of the aldosterone antagonist spironolactone combined with a lower dose of an ACE inhibitor is more effective in reverse left ventricular remodeling in severe congestive heart failure in patients with nonischemic cardiomyopathy.

DETAILED DESCRIPTION:
In the investigators' recent daily clinical practice, they found that the larger dose of the aldosterone antagonist spironolactone combined with a lower dose of an ACE inhibitor and the highest tolerable dose of beta blockers could reverse left ventricular remodeling more effectively than a smaller dose of spironolactone. The ventricular remodeling could get back to normal, especially in patients with none-ischaemic cardiomyopathy. The investigators hypothesize that long term use of a larger dose of the aldosterone antagonist spironolactone could reverse left ventricular remodeling by stimulating new myocyte formation. Thus, they designed this study to verify its efficacy and safety in reversing left ventricular remodeling in severe congestive heart failure in patients with nonischemic cardiomyopathy. To avoid hyperkalemia, the investigators routinely use larger doses of diuretics in combination with a lower dose of an ACE inhibitor to offset the potassium-sparing effects of spironolactone and follow the patients closely.

ELIGIBILITY:
Inclusion Criteria:

* New York Heart Association (NYHA) Functional class Ⅲ or Ⅳ
* Left Ventricular Ejection Fraction (LVEF) <35%
* Nonischemic cardiomyopathy
* Preserved renal function: Cr ≤2.5 mg/dL in males; Cr ≤2.0mg/dL in females

Exclusion Criteria:

* Hyperkalemia (≥5.0 mEg/L)
* Left ventricular systolic dysfunction with pericardial diseases, congenital heart diseases, pulmonary heart diseases, heart valvular diseases, acute coronary syndrome and short life expectancy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2005-09; Study Completion 2009-09 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients whose dilated ventricle reversed to normal (left ventricular end diastolic dimension [LVEDD] defined as <55 mm in males or <50 mm in females and cardiothoracic ratio <50% is normal)

SECONDARY OUTCOMES:
Left ventricular ejection fraction (LVEF)
New York Heart Association (NYHA) functional class
Six-minute walking distance
Cardiogenic death
Cardiac thoracic ratio

CONTACTS AND LOCATIONS:
Overall Officials: Kunshen Liu, M.D., Principal Investigator — The First Hospital of Hebei Medical University
Locations (1):
- The First Hospital of Hebei Medical University, Shijiazhuang, Hebei, China